CLINICAL TRIAL: NCT01500382
Title: A Placebo and Active-Comparator Controlled Multiple-Dose Study to Evaluate the Pharmacokinetics and Pharmacodynamics of MK-4618 in Patients With Overactive Bladder
Brief Title: A Study of the Pharmacokinetics and Pharmacodynamics of Vibegron (MK-4618) in Women With Overactive Bladder (MK-4618-004)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated early due to insufficient recruitment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4618-004
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Overactive Bladder; Overactive Urinary Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide; Tolterodine Tartrate; Chemoprevention; Levofloxacin; Cephalexin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vibegron 100 mg + tolterodine ER 4 mg → placebo (Experimental): During Treatment Period 1, participants will receive 7 days of once-daily vibegron 100 mg and tolterodine extended-release (ER) 4 mg. Participants will then complete a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants will receive 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER.
  Interventions: Drug: Vibegron; Drug: Tolterodine ER; Other: Placebo (vibegron); Other: Placebo (tolterodine ER); Drug: Prophylactic Antibiotic
- Placebo → vibegron 100 mg (Experimental): During Treatment Period 1, participants will receive 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER. Participants will then complete a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants will receive 7 days of once-daily vibegron 100 mg and placebo to match tolterodine ER.
  Interventions: Drug: Vibegron; Other: Placebo (vibegron); Other: Placebo (tolterodine ER); Drug: Prophylactic Antibiotic
- Placebo → tolterodine ER 4 mg (Active Comparator): During Treatment Period 1, participants will receive 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER. Participants will then complete a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants will receive 7 days of once-daily tolterodine 4 mg and placebo to match vibegron.
  Interventions: Drug: Tolterodine ER; Other: Placebo (vibegron); Other: Placebo (tolterodine ER); Drug: Prophylactic Antibiotic
- Placebo → vibegron 50 mg (Experimental): During Treatment Period 1, participants will receive 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER. Participants will then complete a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants will receive 7 days of once-daily vibegron 50 mg and placebo to match tolterodine ER.
  Interventions: Drug: Vibegron; Other: Placebo (vibegron); Other: Placebo (tolterodine ER); Drug: Prophylactic Antibiotic

INTERVENTIONS:
Drug: Vibegron — Tablet, 50 or 100 mg, once daily, for up to 10 days based on treatment assignments and treatment period.
  Other Names: MK-4618
  Arms: Placebo → vibegron 100 mg; Placebo → vibegron 50 mg; Vibegron 100 mg + tolterodine ER 4 mg → placebo
Drug: Tolterodine ER — Capsule, 4 mg, once daily, for up to 10 days based on treatment assignment and treatment period.
  Other Names: Detrol LA™
  Arms: Placebo → tolterodine ER 4 mg; Vibegron 100 mg + tolterodine ER 4 mg → placebo
Other: Placebo (vibegron) — Inactive agent in tablet form, oral administration, once daily, up to 5 weeks, based on treatment assignment in each treatment period.
Other: Placebo (tolterodine ER) — Inactive agent in capsule form, oral administration, once daily, up to 5 weeks, based on treatment assignment in each treatment period.
Drug: Prophylactic Antibiotic — A pre-procedural prophylactic antibiotic (ie, levofloxacin 250 mg, cephalexin) administered orally, 30 minutes prior to each scheduled urodynamic study intervention. It is up to the discretion of the Investigator, based on study protocol recommendations, as to which type of antibiotic may be administered.
  Other Names: Levaquin; Biocef; Ed A-Ceph; Keflex; Keftab; Panixine DisperDose; Zartan

SUMMARY:
The study is designed to investigate the effects of the investigational drug vibegron (MK-4618) compared to placebo on maximum urinary bladder capacity in women with overactive bladder. The study will also evaluate the safety and tolerability of multiple oral doses of vibegron in women with overactive bladder. Overactive bladder is best described as urgency and frequency of urination, with or without involuntary urination and/or the need to awaken during the night to urinate.

The primary efficacy hypothesis is that vibegron is superior to placebo with respect to change from baseline in maximum cystometric capacity at 2 hours postdose on Day 7 (i.e., steady state) in participants with overactive bladder. A true mean increase (vibegron/placebo) of 25% in bladder volume is expected.

The primary safety hypothesis is that administration of multiple oral doses of vibegron is sufficiently well-tolerated in participants with overactive bladder, based on assessment of clinical and laboratory adverse experiences, to permit continued clinical investigation.

DETAILED DESCRIPTION:
Participants will be randomized in each of 2 treatment periods to 1 of 4 possible treatments, which will be administered in double-dummy fashion, and participants will undergo urodynamic procedures prior to dosing on Day 1 and after 7 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-child bearing potential (status post menopausal or post hysterectomy,oophorectomy or tubal ligation). If of reproductive potential, must be non-pregnant (confirmed via blood test) and agree to use (and/or have their partner use) two acceptable methods of birth control beginning at least 2 weeks prior to administration of the first dose of study drug,throughout the study (including washout intervals between treatment periods/panels) and until at least 2 weeks after administration of the last dose of study drug in the last treatment period.
* Body mass index (BMI) of ≤40 kg/m^2 (ie, not morbidly obese)
* Clinical history of overactive bladder symptoms (OAB) for at least 3 months
* Capable of completing an accurate daily diary for reporting purposes

Exclusion Criteria:

* Mentally or legally incapacitated, such as significant emotional problems (other than situational depression) or diagnosed with a significant psychiatric disorder during the past 5-10 years
* Other types of urinary incontinence (ie,stress or mixed)
* History (current or past)of interstitial cystitis, painful bladder syndrome, or chronic pelvic pain or Stage III or greater pelvic organ prolapse
* Other types of kidney/urinary bladder disease/obstruction or infection. Participants with with a history of uncomplicated kidney stones may be enrolled in the study at the discretion of the investigator
* Inability to control bowel movements
* History of narrow angle glaucoma, immunocompromise, stroke, chronic seizures, major neurological disorders and/or other serious and chronic organ-system health conditions (ie, heart disease)
* Urinary catheter, either permanent or intermittent placement
* Failure to meet medication profile requirements or directives required for study eligibility
* Condition for which there is a warning, contraindication, or precaution against the use of tolterodine ER or anticipates the use of prescription medications contraindicated with the use of tolterodine ER
* Daily alcohol or caffeine intake exceeds study requirements (for alcohol: defined as greater than 2 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day; and for caffeine: defined as greater than 3 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee,tea, cola, or other caffeinated beverages (ie, Red Bull) per day
* Inability to refrain from smoking throughout the study's duration
* Illicit drug use
* Recent surgery or recent participation in another clinical trial
* Severe, frequent allergies or history of life-threatening reactions or intolerability to prescription or non prescription medications or food
* Intended or unintended extended absence or exposure to significant change in time zone or sleep schedule (ie, transmeridian travel or shift work) that will interfere with accurate completion of scheduled daily diary entries

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2013-01-02 (Actual); Study Completion 2013-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Vibegron 100 mg + Tolterodine 4 mg → Placebo: During Treatment Period 1, participants received 7 days of once-daily vibegron 100 mg and tolterodine extended-release (ER) 4 mg. Participants then completed a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants received 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER.
- Placebo → Vibegron 100 mg: During Treatment Period 1, participants received 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER. Participants then completed a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants received 7 days of once daily vibegron 100 mg and placebo to match tolterodine ER.
- Placebo → Tolterodine 4 mg: During Treatment Period 1, participants received 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER. Participants then completed a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants received 7 days of once-daily tolterodine 4 mg and placebo to match vibegron.
- Placebo → Vibegron 50 mg: During Treatment Period 1, participants received 7 days of once-daily placebo to match vibegron and placebo to match tolterodine ER. Participants then completed a 2-week single-blind double-dummy placebo washout period prior to Treatment Period 2. During Treatment Period 2, participants received 7 days of once daily vibegron 50 mg and placebo to match tolterodine ER.
Period: Treatment Period 1
Arm/Group | Vibegron 100 mg + Tolterodine 4 mg → Placebo | Placebo → Vibegron 100 mg | Placebo → Tolterodine 4 mg | Placebo → Vibegron 50 mg
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Vibegron 100 mg + Tolterodine 4 mg → Placebo | Placebo → Vibegron 100 mg | Placebo → Tolterodine 4 mg | Placebo → Vibegron 50 mg
Started | 1 | 1 | 1 | 1
Completed | 1 | 1 | 0 | 1
Not Completed | 0 | 0 | 1 | 0
Not completed — Study site went out of business | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Vibegron 100 mg + Tolterodine 4 mg → Placebo | Placebo → Vibegron 100 mg | Placebo → Tolterodine 4 mg | Placebo → Vibegron 50 mg
Started | 1 | 1 | 0 | 1
Completed | 1 | 1 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibegron 100 mg + Tolterodine 4 mg → Placebo | Placebo → Vibegron 100 mg | Placebo → Tolterodine 4 mg | Placebo → Vibegron 50 mg | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (NA) — Only one participant in treatment group. | 61 (NA) — Only one participant in treatment group. | 55 (NA) — Only one participant in treatment group. | 68 (NA) — Only one participant in treatment group. | 58.3 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Fold-change From Baseline in Maximum Cystometric Capacity Post-dose on Day 7
Description: Filling cystometry procedures were performed pre-dose on Day 1 and post-dose on Day 7 in each treatment period. Individual values in fold-change from baseline and post-dose on Day 7 will be natural log-transformed and evaluated with a linear mixed effects model having period and treatment as fixed effects and participant as a random effect.
Time Frame: Baseline (pre-dose Day 1) and Day 7 (post-dose)
Population: Study was terminated by the Sponsor prior to completion. No planned efficacy summaries or analyses were completed.
Groups:
- Vibegron 100 mg: Participants received 7 days of once-daily vibegron 100 mg and placebo to match tolterodine ER 4 mg.
- Vibegron 100 mg + Tolterodine ER 4 mg: Participants received 7 days of once-daily vibegron 100 mg and tolterodine ER 4 mg.
- Vibegron 50 mg: Participants received 7 days of once-daily vibegron 50 mg and placebo to match tolterodine ER 4 mg.
- Placebo: Participants received 7 days of once-daily placebo to match vibegron 100 mg and placebo to match tolterodine ER 4 mg.
Arm/Group | Vibegron 100 mg | Vibegron 100 mg + Tolterodine ER 4 mg | Vibegron 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Fold-change From Baseline in Volume of Urine at First Desire to Void Post-dose on Day 7
Description: as for outcome 1
Time Frame: Baseline (pre-dose Day 1) and Day 7 (post-dose)
Population: Study was terminated by the Sponsor prior to completion. No planned efficacy summaries or analyses were completed.
Arm/Group | Vibegron 100 mg | Vibegron 100 mg + Tolterodine ER 4 mg | Vibegron 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Up to 6 weeks (up to 3 weeks in Period 1 and up to 3 weeks in Period 2)
Population: The All Subjects as Treated (AST) population, which included all participants who received at least one dose of study drug, was used for the safety evaluation. AEs are reported/grouped by drug taken at the time and not by randomly assigned sequence.
Measure: Number; unit: Participants
Arm/Group | Vibegron 100 mg | Vibegron 100 mg + Tolterodine ER 4 mg | Vibegron 50 mg | Placebo
Number analyzed (Participants) | 1 | 1 | 1 | 4
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Discontinued Use of Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. The number of participants who discontinued study drug due to an AE were reported.
Time Frame: Up to 6 weeks (up to 3 weeks in Period 1 and up to 3 weeks in Period 2)
Population: The AST population, which included all participants who received at least one dose of study drug, was used for the safety evaluation. AEs are reported/grouped by drug taken at the time and not by randomly assigned sequence.
Measure: Number; unit: Participants
Arm/Group | Vibegron 100 mg | Vibegron 100 mg + Tolterodine ER 4 mg | Vibegron 50 mg | Placebo
Number analyzed (Participants) | 1 | 1 | 1 | 4
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks (up to 3 weeks in Period 1 and up to 3 weeks in Period 2)
Description: The AST population, which included all participants who received at least one dose of study drug, was used for the safety evaluation. AEs are reported/grouped by drug taken at the time and not by randomly assigned sequence.
Arm/Group | Vibegron 100 mg | Vibegron 100 mg + Tolterodine ER 4 mg | Vibegron 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/4

LIMITATIONS AND CAVEATS:
This study was terminated early due to insufficient recruitment. Only four participants in total participated in the study with three completing and one discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts,or presentations regarding this study 60 days prior to submission for publication/presentation.